CLINICAL TRIAL: NCT05211947
Title: An Open Label, Single Arm, Extension Trial to Examine Long-term Safety of Iclepertin Once Daily in Patients With Schizophrenia Who Have Completed Previous Iclepertin Phase III Trials (CONNEX-X)
Brief Title: A Study to Test Long-term Safety of Iclepertin in People With Schizophrenia Who Took Part in a Previous CONNEX Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision, project discontinued
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0014; 2020-003745-11 (EudraCT Number)
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BI 425809

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with cognitive impairment due to schizophrenia (Experimental)
  Interventions: Drug: BI 425809

INTERVENTIONS:
Drug: BI 425809 — BI 425809
  Other Names: Iclepertin

SUMMARY:
This study is open to adults with schizophrenia who took part in a previous CONNEX study (study 1346-0011, 1346-0012, or 1346-0013). The purpose of this study is to find out how well people with schizophrenia can tolerate a medicine called Iclepertin in the long term.

Participants take Iclepertin as tablets once a day for 1 year. In addition, all participants take their normal medication for schizophrenia.

Participants are in the study for a little more than 1 year. During this time, they visit the study site about 13 times and get about 9 phone calls from the study team.

The doctors collect information on any health problems of the participants. Doctors also regularly check the participants' symptoms of schizophrenia.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent.
* Clinically stable outpatients who have been diagnosed with schizophrenia (as per Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5)).
* Patients, who completed participation in the parent trial.
* Women of childbearing potential must use highly effective methods of birth control.
* Have a study partner who interacts with the patient on a regular basis. Further inclusion criteria apply.

Exclusion criteria:

* Participant who developed DSM-5 diagnosis other than Schizophrenia or any condition that would prevent the patient from participating in the extension trial since enrolment into the parent phase III trial.
* Any suicidal behavior and/or suicidal ideation of type 5 based on the Columbia Suicidality Severity Rating Scale (C-SSRS) in parent trial and up to and including Visit 1 of this study.
* Positive urine drug screen ≥ 3 times during the treatment period of parent trial.
* Patients who are currently or wish to participate in another investigational drug trial.
* Any clinically significant finding or condition in the judgment of the investigator that would jeopardize the patient´s safety while participating in the trial or their capability to participate in the trial.

Further exclusion criteria apply.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1362 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAEs) | up to 1 year and 12 days

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impressions - Severity (CGI-S) to end of treatment (EOT) | up to 1 year
  The CGI-S is a one-item evaluation completed by the clinician on the patient's severity of psychopathology. The CGI-S is rated ordinal from 1 to 7, with 1=normal (not at all ill) to 7=patient among the most extremely ill patients.
Change from baseline in Haemoglobin (Hb) to EOT | up to 1 year

CONTACTS AND LOCATIONS:
Locations (303):
- United States (49):
  - Advanced Research Center, Inc., Anaheim, California
  - Clinical Innovations, Inc, Bellflower, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC (CNS), Garden Grove, California
  - Omega Clinical Trials,LLC, La Habra, California
  - ASCLEPES Research Centers, P.C. dba Alliance Research, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - ATP Clinical Research, Inc., Orange, California
  - NRC Research Institute, Orange, California
  - CNRI - Los Angeles, Pico Rivera, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Velocity Clinical Research-Santa Ana-68902, Santa Ana, California
  - Stanford University Medical Center, Stanford, California
  - Collaborative Neuroscience Research, Torrance, California
  - Institute of Living, Hartford, Connecticut
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Advanced Medical Research Group Inc, Hollywood, Florida
  - Accel Research Sites Network, Maitland, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - CCM Clinical Research Group, LLC-Miami-68482, Miami, Florida
  - Optimus U Corporation-Miami-69452, Miami, Florida
  - University of Miami, Miami, Florida
  - Nova Psychiatry Inc., Orlando, Florida
  - Synexus Clinical Research-Atlanta-67262, Atlanta, Georgia
  - American Medical Research, Chicago, Illinois
  - Sheppard Pratt Physicians's Practice Association, Inc., Baltimore, Maryland
  - Center for Behavioral Health, LLC, Gaithersburg, Maryland
  - PsychCare Consultants Research, St Louis, Missouri
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - Omaha Insomnia and Psychiatric Services, Omaha, Nebraska
  - Hassman Research Institute-Marlton-66897, Marlton, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - New York State Psychiatric Institute, New York, New York
  - Richmond Behavioral Associates-Staten Island-68636, Staten Island, New York
  - UNC Center for Excellence in Community Mental Health, North Carolina Psychiatric Research Center, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Midwest Clinical Research, Dayton, Ohio
  - Insight Clinical Trials, LLC, Independence, Independence, Ohio
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - University of Oregon Prevention Science Institute, Eugene, Oregon
  - Oasis Life Care, State College, Pennsylvania
  - Community Clinical Research, Inc., Austin, Texas
  - Relaro Medical Trials, LLC, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - JPS Center for Behavioral Health Recovery, Fort Worth, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Ben Taub General Hospital, Houston, Texas
  - LinQ Research, LLC-Richmond-70076, Richmond, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (14):
  - Clínica Privada Banfield, Banfield
  - CENYDET-Centro Neurobiologico y de Estres Traumatico (Biopsychomedical Research Group S.R.L.), CABA
  - Fundación para el Estudio y Tratamiento de las Enfermedades Mentales (FETEM), CABA
  - Fundación FunDaMos para la asistencia e investigación en psiquiatría, CABA
  - CEN (Centro Especializado Neurociencias), Córdoba
  - Instituto Modelo de Neurología Lennox, Córdoba
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Sanatorio Morra S.A., Córdoba
  - Instituto de Neurociencias San Agustín, La Plata
  - Global Psy Asociación Civil, La Plata
  - Resolution Psychopharmacology Research Institute, Mendoza
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
  - Centro de Investigacion y Asistencia en Psiquiatria (CIAP), Rosario
  - Centro Medico Luquez, San Vicente
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia
- AKH - Medical University of Vienna, Vienna, Austria
- Belgium (4):
  - CUP Vivalia -La Clairière, Bertix
  - Sint-Kamillus, Bierbeek
  - Universitair Psychiatrisch Centrum Duffel (UPC Duffel), Duffel
  - Meclinas, Mechelen
- Brazil (11):
  - CPN - Centro de Estudos em Neurociências, Belo Horizonte
  - Hospital Sao Jose, Criciúma
  - Trial Tech- Tecnologia em pesquisa com medicamentos, Curitiba
  - J A Serviços Médicos Ltda/ Instituto Goiano de Neuropisquiatria, Goiânia
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
  - Cpquali Pesquisa Clinica Ltda, São Paulo
  - BR Trials, São Paulo
  - Clínica Viver - Centro de Desospitalização Humana, São Paulo
  - Hospital das Clinicas da FMUSP, São Paulo
- Bulgaria (2):
  - Medical Center "Spectar", Plovdiv
  - Filipopolis Ambulatory for Group Practice for Specialized Care in Psychiatry, Plovdiv
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
- Chile (2):
  - Biomedica Research Group, Santiago
  - Psicomed Estudios Clínicos, Segunda Región
- China (23):
  - The sixth People's Hospital of Hebei Province, Baoding
  - Beijing Anding Hospital, Beijing
  - Peking University Sixth Hospital, Beijing
  - Beijing HuiLongGuan Hospital, Beijing
  - The Second People's Hospital of Hunan Province (Brain Hospital of Hunan Province), Changsha
  - The Second Xiangya Hospital Of Central South University, Changsha
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou
  - The third affiliated hospital of Sun Yat-Sen University, Guangzhou
  - Huzhou Third Municipal Hospital, Huzhou
  - Shandong Daizhuang Hospital, Jining
  - The First Affilliated Hospital Of Kunming of Medical College, Kunming
  - Nanjing Brain Hospital, Nanjing
  - The Affilicated Kangning Hospital of Ningbo University, Ningbo
  - Shanghai Mental Health Center, Shanghai
  - Tongji Hospital, Tongji University, Shanghai
  - Shenzhen Kangning Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Anding Hospital, Tianjin
  - Wuxi mental health center, Wuxi
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Xi'an Mental Health Center, Xi'an
  - The Second Affiliated Hospital of Xinxiang Medical Univ., Xinxiang
  - Zhumadian Psychiatric Hospital, Zhumadian
- Colombia (5):
  - Centro de Investigación y Proyectos en neurociencia CIPNA, Barranquilla
  - E.S.E Hospital Mental de Antioquia, Bello
  - Instituto Colombiano del Sistema Nervioso- Clínica Montserrat, Bogotá
  - Centro de Investigaciones del Sistema Nervioso SAS- Grupo Cisne SAS, Bogotá
  - Psynapsis Salud Mental S.A., Pereira
- Croatia (5):
  - Clincal Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Centre Zagreb, Zagreb
  - Solmed Polyclinic, Zagreb
  - Psychiatric Hospital 'Sveti Ivan', Zagreb
  - University Psychiatric Hospital Vrapce, Zagreb
- Czechia (6):
  - National Institute of Mental Health, Klecany
  - MP Meditrine s.r.o., Ostrava
  - A-SHINE s.r.o, Pilsen
  - PRAGTIS s.r.o., Prague
  - INEP medical s.r.o., Prague
  - Psychiatrie Ricany s.r.o., Říčany
- Denmark (3):
  - Aalborg Universitetsshospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Psykiatrisk Center Glostrup, Glostrup Municipality
- Finland (2):
  - Aurora hospital, Helsinki
  - CRST - Clinical Research Services Turku, Turku
- France (8):
  - HOP Charles Perrens, Bordeaux
  - HOP la Colombière, Montpellier
  - HOP Hôtel-Dieu, Nantes
  - HOP Pasteur, Nice
  - HOP Carémeau, Nîmes
  - HOP Guillaume Régnier, Rennes
  - HOP Rouffach, Rouffach
  - HOP Nord-Saint-Priest-en-Jarez-53664, Saint-Priest-en-Jarez
- Germany (9):
  - Zentrum für klinische Forschung Dr. med. I. Schöll GmbH, Bad Homburg
  - Praxis Dr. Hahn, Berlin, Berlin
  - Studienzentrum für Neurologie und Psychiatrie, Böblingen
  - LWL-Klinik Dortmund, Dortmund
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Klinikum der Universität München AÖR, München
  - Universitätsklinikum Tübingen, Tübingen
  - Studienzentrum Nord-West, Westerstede
- Greece (7):
  - Eginition Hospital, Athens
  - Attikon University General Hospital of Attica, Chaïdári
  - Psychiatric Hospital of Attica, Haidari
  - AX Mental Health Clinic, Heraklion
  - General Oncology Hospital "Agioi Anargyri", Nea Kifissia
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Semmelweis University, Budapest, Hungary
- Italy (5):
  - ASST degli Spedali Civili di Brescia, Brescia
  - A.O. Fatebenefratelli, Milan
  - Ist. San Raffaele Turro, Milan
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano (TO)
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (55):
  - Hotei Hospital, Aichi, Konan
  - Okehazama Hospital Fujita Kokoro Care Center, Aichi, Toyoake
  - Toyota Memorial Hospital, Aichi, Toyota
  - National Hospital Organization Shimofusa Psychiatric Medical Center, Chiba, Chiba
  - National Center for Global Health and Medicine Kohnodai Hospital, Chiba, Ichikawa
  - Uematsu Mental Clinic, Fukuoka, Chikugo
  - Mental Clinic Sakurazaka, Fukuoka, Fukuoka
  - AK Clinic, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kuramitsu Hospital, Fukuoka, Fukuoka
  - Hirota Clinic, Fukuoka, Kurume
  - Shiranui Hospital, Fukuoka, Omuta
  - Kishi Hospital, Gumma, Kiryu
  - Obihiro-Kosei General Hospital, Hokkaido, Obihiro
  - Hokudai-dori Mental Health Clinic, Hokkaido, Sapporo
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Tatsuta Clinic, Hyogo, Kobe
  - Kanazawa Medical University Hospital, Ishikwa, Kahoku-gun
  - Kishiro Mental Clinic, Kanagawa, Kawasaki
  - St. Marianna University Hospital, Kanagawa, Kawasaki
  - Links Mental Clinic, Kanagawa, Yokohama
  - Yokohama Onoecho Clinic, Kanagawa, Yokohama
  - Hino Hospital, Kanagawa, Yokohama
  - Yokohama City University Hospital, Kanagawa, Yokohama
  - Kochi Health Sciences Center, Kochi, Kochi
  - Yuge Neuropsychiatric Hospital, Kumamoto, Kumamoto
  - Medical Corporation Yamadakai Yatsushiro Welfare Hospital, Kumamoto, Yatsushiro
  - National Hospital Organization Maizuru Medical Center, Kyoto, Maizuru
  - Tohoku University Hospital, Miyagi, Sendai
  - Shounan Hospital, Nagano, Matsumoto
  - Suwa Red Cross Hospital, Nagano, Suwa
  - Nara Medical University Hospital, Nara, Kashihara
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - University of the Ryukyus Hospital, Okinawa, Ginowan
  - Osaka City Hospital Organization Osaka City General Hospital, Osaka, Osaka
  - National Hospital Organization Hizen Psychiatric Medical Center, Saga, Kanzaki-gun
  - Rainbow and Sea Hospital, Saga, Karatsu
  - Inuo Hospital, Saga, Tosu
  - Nishi Kumagaya Hospital, Saitama, Kumagaya
  - Sho Midori Hospital, Saitama, Saitama
  - Dokkyo Medical University Hospital, Tochigi, Shimotsuga-gun
  - Tokushima University Hospital, Tokushima, Tokushima
  - Medical Corporation Seijin Hospital, Tokyo, Adachi-ku
  - Institute of Science Tokyo Hospital, Tokyo, Bunkyo-ku
  - Nishigahara Hospital, Tokyo, Kita-ku
  - National Center of Neurology and Psychiatry, Tokyo, Kodaira
  - Asuka Hospital, Tokyo, Machida
  - Minami-Aoyama Antique Street Clinic, Tokyo, Minato-ku
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Maynds Tower Mental Clinic, Tokyo, Shibuya-ku
  - Shinjuku East Mental Clinic, Tokyo, Shinjuku-ku
  - Ohwa Mental Clinic, Tokyo, Toshima-ku
  - Hokuriku Hospital, Toyama, Nanto
  - Yamaguchi University Hospital, Yamaguchi, Ube
  - University of Yamanashi Hospital, Yamanashi, Chuo
- Lithuania (4):
  - JSC Romuvos Clinic, Kaunas
  - LUHS KH Psichiatric Clinic Mariu Division, Kaunas
  - JSC Medical center "Puriena", Šilutė
  - Vilnius City Mental Health Center, Vilnius
- Malaysia (4):
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Sentosa, Kuching
  - Hospital Tuanku Ja'afar, Seremban
- Mexico (12):
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Clinica Cemelli, Guadalajara
  - Hospital Aranda de la Parra, León
  - Instituto Nacional de Neurologia y Neurocirugia, Mexico City
  - Centro de Investigación Clinica Acelerada, S.C., Mexico City
  - GabiPros S.C., Mexico City
  - Medical Care & Research SA de CV, Mérida
  - Iecsi S.C., Monterrey
  - CIT-Neuropsique S.C, Monterrey
  - Instituto de Informacion e Investigacion en Salud Mental A.C. (INFOSAME)., Monterrey
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
  - BIND Investigaciones S.C., San Luis Potosí City
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- North Shore Hospital, Takpuna Auckland, New Zealand
- Norway (2):
  - Sykehuset Østfold HF, avd. Moss, Moss
  - Akershus universitetssykehus Oslo, Oslo
- Philippine General Hospital, Manila, Philippines, Philippines
- Poland (9):
  - Psychiatric Doctor's Office Ireneusz Kaczorowski, Bełchatów
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - Health Center Alcea, Gdansk
  - MentalMEDIC, Gliwice
  - Central Teaching Hospital of the Medical University of Lodz, Lodz
  - Individual Specialist Medical Practice Filip Rybakowski, Poznan
  - EUROMEDIS Sp. z o.o., Szczecin, Szczecin
  - Institute of Psychiatry and Neurology in Warsaw, Warsaw
  - Clinhouse, Zabrze
- ULS da Região de Leiria, E.P.E., Leiria, Portugal
- Romania (2):
  - Mental Health Center Sector 4, Bucharest
  - SC Carpe Diem SRL, Sibiu
- Serbia (6):
  - Clinical Hospital Center Dr. Dragisa Misovic, Belgrade
  - General Hospital Euromedik, Belgrade
  - Institute for Mental Health, Belgrade
  - Special Hospital for Psychiatric Diseases Gornja Toponica, Gornja Toponica
  - Special Hospital for Psychiatric Diseases Sveti Vračevi, Novi Kneževac
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (3):
  - Psychiatria, Nemocnica s poliklinikou Prievidza so sidlom v Bojniciach, Bojnice
  - EPAMED s.r.o., Košice
  - Psychiatricka Ambulancia Psycholine s.r.o., Rimavská Sobota
- South Korea (8):
  - Inje University Busan Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (10):
  - Hestia Palau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario General de Villalba, Collado de Villalba
  - Hospital Universitario Reina Sofía-Córdoba-40500, Córdoba
  - Hospital Puerta de Hierro, Majadahonda
  - Centro de Salud de San Juan, Salamanca
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico de Valencia, Valencia
  - Hospital Nicolás Peña, Vigo
  - Hospital Provincial. Complejo Asistencial de Zamora, Zamora
- Sweden (2):
  - Psykiatriska Kliniken, Helsingborg
  - Akademiska sjukhuset, Uppsala
- Taiwan (8):
  - Kai-Syuan Psychiatric Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Keelung, Keelung
  - Chung Shan Medical University Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taoyuan Psychiatric Center, Taoyuan District
  - Chang Gung Memorial Hospital(Linkou), Taoyuan District
- Turkey (Türkiye) (5):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara University Medical School, Ankara
  - Istanbul University, Istanbul
  - Dokuz Eylul Universitesi Psikiyatri A.B.D., Izmir
  - Celal Bayar Universitesi Tip Fakultesi, Manisa
- Communal Non-Profit Enterprise "Regional Clinical Psychiatric Hospital" of Kirovohrad Regional Council, Nove, Ukraine
- United Kingdom (8):
  - Bodmin Community Hospital, Bodmin
  - The Fritchie Centre, Cheltenham
  - Redesmere, Chester
  - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Maudsley Hospital, London
  - Warneford Hospital, Oxford
  - Moorgreen Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com